CLINICAL TRIAL: NCT02015754
Title: Irinotecan -Eluting LC Bead-M1 (DEBIRI-M1) for Patients With Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1305; NA_00078095 [JHMIRB]
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DEBIRI (Experimental)
  Interventions: Drug: DEBIRI; Device: LC Bead M1; Procedure: TACE

INTERVENTIONS:
Drug: DEBIRI — Irinotecan hydrochloride is a semisynthetic derivative of camptothecin, an alkaloid extracted from the tree Camptotheca acuminata. Irinotecan hydrochloride trihydrate is a pale yellow to yellow crystalline powder, it is mixed in DC Beads and injected in the tumor.
Device: LC Bead M1 — The LC Bead M1, loaded with irinotecan (DEBIRI-M1) to treat patients with hepatic metastases from colorectal cancer.
Procedure: TACE — TACE a minimally invasive procedure performed to restrict a tumor's blood supply.

SUMMARY:
Purpose:

The purpose of this study is to determine the feasibility and safety of using small beads (70-150 micron in place of 100-300 micron) to deliver chemotherapy into the liver to treat patients with liver lesions from colorectal cancer. The beads (LC-Bead M1) will be loaded with irinotecan (DEBIRI-M1), and used to administer transarterial chemoembolization (TACE).

Eligibility:

Patients with liver cancer from colorectal cancer.

Study Overview/ Treatment:

DEBIRI, loaded with irinotecan, is a device that utilizes tiny beads (70-150 microns) to deliver chemotherapy agents into liver tumor(s) via the hepatic artery. This device allows for continuous release of irinotecan into the liver tumor tissue(s) causing necrosis of the targeted tumor(s). The potential advantages of the smaller beads are deeper penetration into the tumor bed, while avoiding premature proximal occlusion of vessels feeding the tumor, and more consistent dosing. Response to therapy will be evaluated monthly by clinic visits and blood tests (to include assessment of liver function and tumor markers) and by imaging (usually MRIs) every 1-2 months. Patients will be on study for 6 months after which they will be exited from the study and followed for survival. Once exited from the study they will continue to be eligible to receive DEBIRI, should it be recommended.

ELIGIBILITY:
Inclusion Criteria:

-Patients with a diagnosis of colorectal cancer with hepatic metastases who have failed or are intolerant to at least one systemic chemotherapy or liver directed therapy.

1. The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at study entry.
2. The patient is age 18 years or older.
3. The patient has a life expectancy of >12 weeks.
4. Patients with liver dominant disease defined as >/=75% tumor body burden confined to the liver
5. Less than 60% liver tumor replacement
6. At least one month has elapsed since most recent prior cancer therapy with the following exception:

   -Chemotherapy (excluding irinotecan based regimens) may continue if there is evidence of hepatic progression on treatment providing there is no change in the therapy in the 1 month prior to DEBIRI-TACE treatment and any immediate chemotherapeutic toxicity that will complicate DEBIRI-TACE is resolved. In this case, the chemotherapy may continue because it is continuing to control the extrahepatic disease.
7. The patient has measurable disease that will be directly treated with intrahepatic therapy (as defined by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).
8. Patients with at least one measurable liver metastases> 2 cm.
9. Patients with patent main portal vein
10. The patient has adequate hematologic function as defined by the following criteria:

    -An absolute neutrophil count (ANC) >/= 1500/mL, Hemoglobin >/= 9.5 g/dL, and a Platelet count >/=75,000/mL, INR </=1.3 prior to receiving DEBIRI-TACE.
11. The patient has adequate hepatic function, as defined by the following criteria:

    -Total bilirubin</= 2.0 mg/dL, Aspartate transaminase (AST) and alanine transaminase (ALT) </= 5 x the upper limit of normal (ULN), Albumin >2.
12. The patient has adequate renal function, as defined by the following criteria:

    -Serum creatinine</=2.0.
13. The patient has a baseline international normalized ratio (INR)<1.5.
14. The patient, if a woman of childbearing potential, has a negative pregnancy test.
15. The patient is able to give written informed consent.
16. The patient is willing and able to comply with study procedures, scheduled visits, and treatment plans.

Exclusion Criteria:

1. The patient has a history of another primary cancer (ie, a primary cancer not associated with the patient's current liver tumor), with the exception of (a) curatively resected nonmelanomatous skin cancer; (b) curatively treated cervical carcinoma in situ; or (c) other primary solid tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years prior to enrollment (date of informed consent).
2. Any contraindication for hepatic embolization procedures:

   * Large shunt as determined by the investigator (pretesting with TcMMA not required)
   * Severe atheromatosis
   * Hepatofugal blood flow
   * Main portal vein occlusion (e.g. thrombus or tumor)
   * Any patient eligible for curative treatment (i.e. resection or radiofrequency ablation)
   * Patients' whose only measurable disease is within an area of the liver previously subject to radiotherapy
3. Contraindications to irinotecan:

   * Chronic inflammatory bowel disease and/or bowel obstruction
   * History of severe hypersensitivity reactions to irinotecan hydrochloride trihydrate, lactic acid or to any of the excipients of Camptosar
   * Severe bone marrow failure
   * History of Gilbert Syndrome (specific testing not required)
   * Concomitant use with St John's Wort (Hypericum)
   * Marco-shunting noted on the hepatic angiogram.
4. The patient has untreatable bleeding diathesis.
5. The patient has complete main portal vein thrombosis with reversal of flow.
6. The patient has evidence of clinically significant peripheral vascular disease.
7. The patient has brain metastases
8. The patient has clinically significant or symptomatic extrahepatic disease, for example, an uncontrolled intercurrent illness including, but not limited to:

   * Ongoing or active infection requiring parenteral antibiotics
   * Symptomatic congestive heart failure (class II to IV of the New York Heart Association classification for heart disease)
   * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
   * Uncontrolled hypertension (systolic blood pressure>150 mmHg, diastolic blood pressure>90 mmHg, found on 2 consecutive measurements separated by a 1-week period despite adequate medical support)
   * Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [NCI-CTCAE Grade 3] or asymptomatic sustained ventricular tachycardia)
9. The patient is pregnant or breast-feeding.
10. Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements
11. There is evidence of substance abuse or medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results
12. The patient is allergic to contrast media that cannot be readily prevented with premedication or managed.
13. Other significant medical or surgical condition, or any medication or treatment, that would place the patient at undue risk and that would preclude the safe use of chemoembolization or would interfere with study participation
14. The patient has peritoneal disease or ascites (greater than trace on imaging).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2016-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.F. Geschwind, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients diagnosed with colorectal cancer with unresectable hepatic metastases who have failed or were intolerant to at least one line of systemic chemotherapy or liver-directed therapy. Patients were enrolled at Johns Hopkins to receive transarterial chemoembolization (TACE) therapy. The last patient completed in June 2015.
Period: Overall Study
Arm/Group | DEBIRI
Started | 14 (17 participants were consented, but 3 participants were screened out prior to treatment)
Completed First TACE (Number of patients who completed the first treatment on protocol and included in analysis.) | 14
Completed First Clinical and Imaging (Participants completing this milestone will be analyzed for image response outcomes) | 13 (1 patient exited prior to follow-up)
Completed (Participants who have completed all 24 weeks of treatment on trial) | 3
Not Completed | 11
Not completed — Disease progression | 5
Not completed — Change in treatment modality | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | DEBIRI
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 52.5 [44 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Out of 14 enrolled participants, 10 participants identified as non-Hispanic and 4 patients did not elect to reveal their ethnicity.
  From the 14 participants, 9 were white, 4 were black or African American, and 1 was unknown.
  Participants
    Non-Hispanic: number analyzed (Participants) | 10
    Non-Hispanic: White | 6
    Non-Hispanic: Black or African American | 4
    Non-Hispanic: Unknown | 0
    Unknown: number analyzed (Participants) | 4
    Unknown: White | 3
    Unknown: Black or African American | 0
    Unknown: Unknown | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Success of DEBIRI-M1 Procedure as a Measure of Feasibility (Percentage of Successful Treatments)
Description: Feasibility is defined as achieving an acceptable level of technical success in the use of DEBIRI beads treating hepatic metastases in patients with colorectal cancer.
Time Frame: 6 months
Population: The 14 patients received a total of 32 DEBIRI-M1 TACE procedures.
Measure: Number; unit: percentage of successful treatments
Units Other Than Participants: DEBIRI-M1 Treatments
Arm/Group | DEBIRI
Number analyzed (Participants) | 14
Number analyzed (DEBIRI-M1 Treatments) | 32
percentage of successful treatments | 100

2. Primary Outcome: Safety, Defined as Demonstrating Tolerable Device-related Toxicity Profile in the Use of DEBIRI Beads Used to Treat Hepatic Metastases in Patients With Colorectal Cancer
Description: Toxicities assessed as being at least possibly related will be recorded including system organ class, subclass, grade, frequency and time interval from DEBIRI-M1.
Time Frame: 6 weeks
Population: 6-week toxicity report of device-related adverse events for all 14 participants. Classification and grading based on CTCAE v4.0.
Measure: Count of Participants; unit: Participants
Arm/Group | DEBIRI
Number analyzed (Participants) | 14
Participants
  Grade 1-2 Adverse Events: Elevated ALP | 2
  Grade 1-2 Adverse Events: Hypoalbuminemia | 1
  Grade 1-2 Adverse Events: Abdominal pain | 3
  Grade 1-2 Adverse Events: Anemia | 2
  Grade 1-2 Adverse Events: Nausea | 1
  Grade 1-2 Adverse Events: Leukopenia | 1
  Grade 1-2 Adverse Events: 30-day mortality | 0
  Grade 1-2 Adverse Events: Participants with no events | 4
  Grade 3-4 Adverse Events: Elevated ALP | 0
  Grade 3-4 Adverse Events: Hypoalbuminemia | 0
  Grade 3-4 Adverse Events: Abdominal pain | 4
  Grade 3-4 Adverse Events: Anemia | 0
  Grade 3-4 Adverse Events: Nausea | 0
  Grade 3-4 Adverse Events: Leukopenia | 0
  Grade 3-4 Adverse Events: 30-day mortality | 0
  Grade 3-4 Adverse Events: Participants with no events | 10

3. Secondary Outcome: Efficacy - Tumor Response by RECIST
Description: Efficacy as assessed by radiographic tumor response using the RECIST criteria at baseline and at 6-week imaging following TACE treatments.
  Complete Response (CR): Disappearance of all lesions targeted by DEBIRI-M1 Partial Response (PR): At least 30% decrease in sum of longest diameter (LD) of lesions targeted by DEBIRI-M1, taking as reference the baseline sum LD Progressive Disease (PD): At least 20% increase in sum of the LD Of lesions targeted by DEBIRI-M1, taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, of lesions targeted by DEBIRI-M1, taking as reference the smallest sum LD since treatment started
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DEBIRI
Number analyzed (Participants) | 13
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 8
  Progressive Disease | 4
  Objective response (CR + PR) | 1
  Disease control rate (CR + PR + SD) | 9

4. Secondary Outcome: Efficacy - Tumor Response by mRECIST
Description: Efficacy as assessed by radiographic tumor response using modified RECIST (mRECIST) criteria at baseline and at 6-week imaging following TACE treatments.
  Complete Response (CR): Disappearance of any intratumoral arterial enhancement in all target lesions Partial Response (PR): At least 30% decrease in the sum of diameters of viable target lesions, taking as reference the baseline sum of the diameters of target lesions Progressive Disease (PD): At least 20% increase in sum of diameters of viable target lesions, taking as reference the smallest sum of diameters of viable target lesions since treatment started.
  Stable Disease (SD): Any cases that do not qualify for either PR or PD.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DEBIRI
Number analyzed (Participants) | 13
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 9
  Progressive Disease | 4
  Objective response (CR + PR) | 0
  Disease control rate (CR + PR + SD) | 9

5. Secondary Outcome: Efficacy -Tumor Response by European Association for the Study of the Liver (EASL) Criteria
Description: Efficacy as assessed by radiographic tumor response using EASL amendment at baseline and at 6-week imaging following TACE treatments.
  Complete Response (CR): Achieving 100% tumor necrosis of lesions targeted by DEBIRI-M1. Baseline degree of tumor enhancement used as a reference.
  Partial Response (PR): Demonstrating greater than 50% tumor necrosis in lesions targeted by DEBIRI-M1.
  Stable Disease (SD): Not meeting requirements for CR or PR and not demonstrating evidence of progression of lesions targeted by DEBIRI-M1.
  Progressive Disease (PD): Reappearance of or increased tumor enhancement greater than 25% in lesions previously targeted by DEBIRI-M1.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DEBIRI
Number analyzed (Participants) | 13
Participants
  Complete Response | 0
  Partial Response | 3
  Stable Disease | 4
  Progressive Disease | 6
  Objective response (CR + PR) | 3
  Disease control rate (CR + PR + SD) | 7

6. Secondary Outcome: Efficacy - Tumor Response by World Health Organization (WHO) Criteria
Description: Efficacy as assessed by radiographic tumor response using WHO criteria at baseline and at 6-week imaging following TACE treatments.
  Complete Response (CR): No lesions detected for at least 4 weeks. Partial Response (PR): 50% or greater decrease in the sum of the products of diameters Stable Disease (SD): Cases that do not fit the criteria of PR or PD. Progressive Disease (PD): 25% or greater increase in the sum of the products of diameters in one or more lesions; or new lesions
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DEBIRI
Number analyzed (Participants) | 13
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 9
  Progressive Disease | 3
  Objective response (CR + PR) | 1
  Disease control rate (CR + PR + SD) | 10

7. Secondary Outcome: Number of Participants With Change in Carcinoembryonic Antigen (CEA)
Description: CEA measurements pre- and post- DEBIRI treatment will be recorded to ascertain if it is predictive of survival.
Time Frame: 6 weeks
Population: 2 out of original 14 patients had no CEA measurements.
Measure: Number; unit: participants
Arm/Group | DEBIRI
Number analyzed (Participants) | 12
participants | 6
Statistical Analysis 1: Comparison: DEBIRI; Multivariate Cox-regression analysis to identify independent prognostic factors for overall survival from baseline characteristics. Relative risk with 95% confidence intervals calculated as measure of association; Test type: Other; p = 0.004, Regression, Cox — Differences of p-value < 0.05 considered statistically significant

8. Secondary Outcome: Median Overall Survival
Description: Median overall survival from start of therapy (DEBIRI #1) until death (or date of censor).
Time Frame: Up to 26 months
Measure: Median (Full Range); unit: months
Arm/Group | DEBIRI
Number analyzed (Participants) | 14
months | 18.7 [1.1 to 25.83]

9. Secondary Outcome: One-year Survival Percentage
Description: Percentage of study patients surviving after one year from initial treatment analyzed with Kaplan-Meier curve.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | DEBIRI
Number analyzed (Participants) | 14
percentage of participants | 36

10. Other Pre Specified Outcome: Exploratory Endpoint - Pharmacokinetic (PK) Profile of Irinotecan and SN-38 Post DEBIRI-TACE
Description: PK analysis of irinotecan and its metabolite SN-38 in the first 10 patients enrolled on protocol including peak plasma concentration (Cmax). Time points assessed in protocol were pre-dose, and then 5min, 10min, 15min, 30min, 1hr, 2hr, 4hr, 6hr, and 24hr post administration of 100mg irinotecan.
Time Frame: 24 hours
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | DEBIRI
Number analyzed (Participants) | 10
ng/mL
  Cmax irinotecan | 1299 (2276)
  Cmax SN-38 | 41.5 (26.1)

11. Other Pre Specified Outcome: Exploratory Endpoint -Total Drug Exposure Over Time (AUC) of Irinotecan and SN-38 Post DEBIRI-TACE
Description: Total drug exposure over time (AUC) of irinotecan and its metabolite SN-38 post DEBIRI-TACE in the first 10 patients enrolled on protocol. Time points assessed in protocol were pre-dose, and then 5min, 10min, 15min, 30min, 1hr, 2hr, 4hr, 6hr, and 24hr post administration of 100mg irinotecan.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DEBIRI
Number analyzed (Participants) | 10
ng*h/mL
  AUC irinotecan | 5020 (2138)
  AUC SN-38 | 305 (206)

12. Other Pre Specified Outcome: Exploratory Endpoint -Tmax of Irinotecan and SN-38 Post DEBIRI-TACE
Description: Time taken to reach maximum concentration (Tmax) of irinotecan and its metabolite SN-38 post DEBIRI-TACE in the first 10 patients enrolled on protocol. Time points assessed in protocol were pre-dose, and then 5min, 10min, 15min, 30min, 1hr, 2hr, 4hr, 6hr, and 24hr post administration of 100mg irinotecan.
Time Frame: 24 hours
Measure: Median (Standard Deviation); unit: hours
Arm/Group | DEBIRI
Number analyzed (Participants) | 10
hours
  Tmax of irinotecan | .95 (.77)
  Tmax of SN-38 | 1.26 (.54)

13. Other Pre Specified Outcome: Plasma Half-life of Irinotecan and SN-38 Post DEBIRI-TACE
Description: Plasma half-life (t 1/2) of irinotecan and its metabolite SN-38 post DEBIRI-TACE in the first 10 patients enrolled on protocol. Time points assessed in protocol were pre-dose, and then 5min, 10min, 15min, 30min, 1hr, 2hr, 4hr, 6hr, and 24hr post administration of 100mg irinotecan.
Time Frame: 24 hours
Measure: Median (Standard Deviation); unit: hours
Arm/Group | DEBIRI
Number analyzed (Participants) | 10
hours
  t 1/2 irinotecan | 5.7 (1.2)
  t 1/2 SN-38 | 8.6 (2.6)

14. Other Pre Specified Outcome: Exploratory Endpoint - Angiogenesis
Description: Changes in vascular endothelial growth factors (VEGF), VEGF receptors VEGFR1 and VEGFR2 pre- and post- DEBIRI treatment examined for significant effects as well as association with DEBIRI treatment. One-sample Wilcoxon signed rank test was utilized to compare whether %change of VEGF, VEGFR1, or VEGFR2 from baseline was equal to 0. For groups with non-zero percent changes, the 95% confidence intervals were provided.
Time Frame: 24 hours
Measure: Median (95% Confidence Interval); unit: % change from baseline
Arm/Group | DEBIRI
Number analyzed (Participants) | 14
% change from baseline
  VEGF (immediately post) | -2.66 [-19.5 to 6.45]
  VEGF (24 hours post) | 6.37 [-6.03 to 43.0]
  VEGFR1 (immediately post) | 4.02 [-13.7 to 19.8]
  VEGFR1 (24 hours post) | -37.9 [-45.6 to -19.6]
  VEGFR2 (immediately post) | 4.49 [-2.07 to 11.2]
  VEGFR2 (24 hours post) | 5.51 [-5.24 to 18.7]
Statistical Analysis 1: Comparison: DEBIRI; Test type: Other — VEGF immediately post treatment; p = 0.6257, one-sample Wilcoxon signed rank test
Statistical Analysis 2: Comparison: DEBIRI; Test type: Other — VEGF at 24 hours post treatment; p = 0.4143, one-sample Wilcoxon signed rank test
Statistical Analysis 3: Comparison: DEBIRI; Test type: Other — VEGFR1 immediately post treatment; p = 0.583, one-sample Wilcoxon signed rank test
Statistical Analysis 4: Comparison: DEBIRI; Test type: Other — VEGFR1 at 24 hours post treatment; p = .0012, one-sample Wilcoxon signed rank test
Statistical Analysis 5: Comparison: DEBIRI; Test type: Other — VEGFR2 immediately post treatment; p = 0.1353, one-sample Wilcoxon signed rank test
Statistical Analysis 6: Comparison: DEBIRI; Test type: Other — VEGFR2 at 24 hours post treatment; p = 0.2163, one-sample Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: Adverse events collected through study completion, an average of 6 months.
Arm/Group | DEBIRI
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEBIRI (N=14)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEBIRI (N=14)
Abdominal pain (Gastrointestinal disorders) | 11 (12)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 6 (7)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 2 (2)
INR increased (Investigations) | 3 (3)
Fatigue (General disorders) | 8 (12)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
White blood cell decreased (Investigations) | 2 (4)
Lymphocyte count decreased (Investigations) | 5 (7)
Nausea (Gastrointestinal disorders) | 4 (6)
Neutrophil count decreased (Investigations) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Platelet count decreased (Investigations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No